CLINICAL TRIAL: NCT06963073
Title: Effect of Education and Tele-Follow-Up Program Given to New Type 2 Diabetes Patients on Diabetes Self-Management and Blood Glucose Regulation
Brief Title: The Effect of Education and Tele-Follow-Up Program on Diabetes Self-Management and Blood Glucose Regulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Naile ALANKAYA, Associate Professor, PhD, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COMU-SBF-NA-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Self-Management; Blood Glucose Regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: In the research, firstly, a pre-test (Introductory Information Form, "Adult Diabetes Knowledge Scale" to assess their knowledge about the disease, and the "Diabetes Self-Management Scale) will be applied to intervention and control groups. Blood glucose levels and Hemoglobin A1c (HbA1c) values will be obtained from the patients' hospital records on the day of measurement. In the randomized experimental group, participants will receive one-on-one face-to-face diabetes education. Participants in the control group will receive only the educational booklet prepared by the researcher, without any formal education. Participants who attended the training will be contacted by phone at least three times-two weeks, one month, and two months after the training. After the applications are completed, a posttest.If available, fasting blood glucose and Hemoglobin A1c values will be obtained from the hospital records on the corresponding date.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic DM (Experimental): The intervention group will consist of 30 people. This group will be given 45 minutes of diabetes education (nutrition, exercise, medication, treatment, insulin administration, etc.).
  Interventions: Other: Diabetic DM
- Control group (No Intervention): The control group will consist of 30 people. No training will be given to this group. Only a brochure containing brief diabetes information will be given.

INTERVENTIONS:
Other: Diabetic DM — The intervention group will receive 45 minutes of diabetes education. Three telemonitoring sessions will be held 2 weeks, 1 month and 3 months after the education. During the monitoring, participants will be asked to monitor their blood sugar and HbA1C values, if any. Nothing will be done to the control group. The same monitoring will be held for the control group 3 months later.
  Other Names: Diabetes training
  Arms: Diabetic DM

SUMMARY:
This study is designed as a randomized controlled trial to determine the effects of education and the Tele-Follow-up program on the disease knowledge, self-management, and blood glucose regulation of newly diagnosed Type 2 diabetes patients.

DETAILED DESCRIPTION:
The population for this study consists of newly diagnosed Type 2 diabetes patients who visit the Dr. Burhan Nalbantoğlu Hospital. This study was planned as a randomized controlled trial. In the study, simple randomization design was preferred among experimental designs. Computer-generated random numbers method was used in sample size calculation. The sample size was calculated using the "G. Power-3.1.9.2" program, and the minimum required sample size for the study was determined before data collection at a 95% confidence level. According to the calculation, for the independent sample t-test with a 0.05 alpha value, a 1.128 effect size, and a theoretical power of 95%, the minimum sample size was determined to be 44 participants (22 per group). By considering that there might be losses in the study, it is planned to include a total of 60 patient in the study.

Data collection will take place in three stages.

1. All participants eligible for the study (both experimental and control groups) will be required to complete the "Demographic Information Form," the "Adult Diabetes Knowledge Scale" to assess their knowledge about the disease, and the "Diabetes Self-Management Scale" to evaluate their diabetes self-management. Blood glucose levels and Hemoglobin A1c (HbA1c) values will be obtained from the patients' hospital records on the day of measurement. For Body Mass Index (BMI), the researcher will measure the patients' height and weight, and BMI will be calculated. In the randomized experimental group, participants will receive one-on-one face-to-face diabetes education in a dedicated training room, delivered via a PowerPoint presentation prepared by the researcher, using a computer. At the end of the training, an educational booklet will be provided. Participants in the control group will receive only the educational booklet prepared by the researcher, without any formal education. After three months, participants in the control group will be informed that they will receive individual education at the end of the study.
2. Participants who attended the training will be contacted by phone at least three times-two weeks, one month, and two months after the training. The effects of the education on diabetes management will be evaluated, home-monitored blood glucose levels will be inquired and recorded, and additional education will be provided where necessary.
3. Three months after the initial planned education and following telemonitoring (after at least three follow-up phone calls), the "Adult Diabetes Knowledge Scale" and the "Diabetes Self-Management Scale" will be re-administered by the patients in order to evaluate the impact of the education on diabetes management. If available, fasting blood glucose and Hemoglobin A1c values will be obtained from the hospital records on the corresponding date. Participants in the control group will also be asked to complete the same questionnaires again. After the data collection process is completed, the same planned education will be provided to participants in the control group as well, in order to eliminate any potential disadvantage or ethical concerns.

The data collection tools to be used in this study include the Descriptive Characteristics Form, the Adult Diabetes Knowledge Scale, and the Diabetes Self-Management Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study.
2. Having recently been diagnosed with Type 2 Diabetes.
3. Not having cognitive dysfunction.
4. Not having done diabetes education before.

Exclusion Criteria:

1. Being under 18 years of age.
2. Having cognitive dysfunction.
3. Not volunteering to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management Scale | Baseline and after 6 months
  As a result of the study by Koç and his colleagues, a new measurement tool called "Type 2 Diabetes Self-Management Scale" was developed. A minimum of 19 and a maximum of 95 points can be obtained from the scale. There is no cut-off score range for the scale. According to the total score average, high scores indicate good self-management, while low scores indicate poor self-management.
Adult Diabetes Knowledge Scale | Baseline and after 6 months
  The scale was developed by Erener Yavuz and Erol (2019) to measure the knowledge levels of adult diabetic individuals. The maximum score that can be obtained from the scale is 28, and the minimum score is 0. Scores between 14 and 28 indicate a high level of knowledge, while scores below 14 indicate insufficient level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: NAİLE ALANKAYA, Assosiate Prof., Study Director — Çanakkale Onsekiz Mart University, Faculty of Health Sciences
Locations (2):
- Turkey (Türkiye) (2):
  - Çanakkale Onsekiz Mart University, Faculty of Health Sciences, Çanakkale
  - Çanakkale Onsekiz Mart University, Faculty of Health Sciences, Çanakkale, Çanakkale

IPD SHARING:
Plan to Share IPD: No